CLINICAL TRIAL: NCT05765760
Title: Improvement of Acute Respiratory Distress Syndrome Ventilation-perfusion Matching by Prone Positioning Assessed by Electrical Impedance Tomography
Brief Title: Improvement of ARDS Ventilation-perfusion Matching by Prone Positioning Assessed by EIT
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Rui Wang, Principal Investigator, Beijing Chao Yang Hospital
Other Study IDs: 2022-KE-615
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Respiratory Distress Syndrome; Prone Position; Electrical Impedance Tomography
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood gas analysis, blood routine, liver and kidney function, coagulation, and BNP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a highly lethal disease with limited treatment options. In recent years, prone position ventilation has been shown to improve the mortality rate and lung injury of ARDS patients by promoting lung recruitment, improving ventilation/perfusion (V/Q) ratio, enhancing respiratory system compliance, promoting sputum drainage, and effectively avoiding overinflation of the dorsal lung. Electrical Impedance Tomography (EIT) technology has been used to evaluate the effect of prone position ventilation on lung V/Q matching, and some studies have confirmed that prone position ventilation can improve lung V/Q matching and oxygenation index. However, previous studies were mostly case reports or small-sample physiological studies that lacked dynamic changes in lung V/Q matching during repeated prone position ventilation. Therefore, this study hypothesizes that prone position ventilation can increase lung V/Q matching in ARDS patients, and its improvement is correlated with changes in oxygenation index, invasive ventilation time, and patient prognosis. Repeated prone position ventilation can maintain lung V/Q matching at a higher level, no longer affected by changes in body position, which can accelerate pulmonary function recovery and improve the prognosis of ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. meet the diagnostic criteria of Berlin's definition for ARDS;
3. invasive ventilation time < 48h;
4. PaO2/FiO2 < 150mmHg.

Exclusion Criteria:

1. Contraindication to the prone position;
2. Contraindication to the EIT;
3. Hemodynamically unstable;
4. Patients with hypernatremia;
5. Patients have received extracorporeal membrane oxygenation treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ARDS Patients with PaO2/FiO2 < 150mmH
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
ICU mortality | 28 days after enrollment
  The death of patients that occurs during their stay in the ICU

SECONDARY OUTCOMES:
Ventilator-free days | 28 days after enrollment
  Days without receiving invasive ventilation at day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Wang, Dr., Study Director — Beijing Chao-Yang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Attaway AH, Scheraga RG, Bhimraj A, Biehl M, Hatipoglu U. Severe covid-19 pneumonia: pathogenesis and clinical management. BMJ. 2021 Mar 10;372:n436. doi: 10.1136/bmj.n436. PMID 33692022
- [Background] Slobod D, Damia A, Leali M, Spinelli E, Mauri T. Pathophysiology and Clinical Meaning of Ventilation-Perfusion Mismatch in the Acute Respiratory Distress Syndrome. Biology (Basel). 2022 Dec 30;12(1):67. doi: 10.3390/biology12010067. PMID 36671759
- [Background] Borges JB, Costa EL, Bergquist M, Lucchetta L, Widstrom C, Maripuu E, Suarez-Sipmann F, Larsson A, Amato MB, Hedenstierna G. Lung inflammation persists after 27 hours of protective Acute Respiratory Distress Syndrome Network Strategy and is concentrated in the nondependent lung. Crit Care Med. 2015 May;43(5):e123-32. doi: 10.1097/CCM.0000000000000926. PMID 25746507
- [Background] Borges JB, Hansen T, Larsson A, Hedenstierna G. The "normal" ventilated airspaces suffer the most damaging effects of mechanical ventilation. Intensive Care Med. 2017 Jul;43(7):1057-1058. doi: 10.1007/s00134-017-4708-1. Epub 2017 Feb 15. No abstract available. PMID 28204859
- [Background] Terragni PP, Rosboch G, Tealdi A, Corno E, Menaldo E, Davini O, Gandini G, Herrmann P, Mascia L, Quintel M, Slutsky AS, Gattinoni L, Ranieri VM. Tidal hyperinflation during low tidal volume ventilation in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2007 Jan 15;175(2):160-6. doi: 10.1164/rccm.200607-915OC. Epub 2006 Oct 12. PMID 17038660
- [Background] Rampon GL, Simpson SQ, Agrawal R. Prone Positioning for Acute Hypoxemic Respiratory Failure and ARDS: A Review. Chest. 2023 Feb;163(2):332-340. doi: 10.1016/j.chest.2022.09.020. Epub 2022 Sep 23. PMID 36162482
- [Background] Gattinoni L, Taccone P, Carlesso E, Marini JJ. Prone position in acute respiratory distress syndrome. Rationale, indications, and limits. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1286-93. doi: 10.1164/rccm.201308-1532CI. PMID 24134414
- [Background] Fernandez R, Trenchs X, Klamburg J, Castedo J, Serrano JM, Besso G, Tirapu JP, Santos A, Mas A, Parraga M, Jubert P, Frutos F, Anon JM, Garcia M, Rodriguez F, Yebenes JC, Lopez MJ. Prone positioning in acute respiratory distress syndrome: a multicenter randomized clinical trial. Intensive Care Med. 2008 Aug;34(8):1487-91. doi: 10.1007/s00134-008-1119-3. Epub 2008 Apr 22. PMID 18427774
- [Background] Taccone P, Pesenti A, Latini R, Polli F, Vagginelli F, Mietto C, Caspani L, Raimondi F, Bordone G, Iapichino G, Mancebo J, Guerin C, Ayzac L, Blanch L, Fumagalli R, Tognoni G, Gattinoni L; Prone-Supine II Study Group. Prone positioning in patients with moderate and severe acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2009 Nov 11;302(18):1977-84. doi: 10.1001/jama.2009.1614. PMID 19903918
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Mathews KS, Soh H, Shaefi S, Wang W, Bose S, Coca S, Gupta S, Hayek SS, Srivastava A, Brenner SK, Radbel J, Green A, Sutherland A, Leonberg-Yoo A, Shehata A, Schenck EJ, Short SAP, Hernan MA, Chan L, Leaf DE; STOP-COVID Investigators. Prone Positioning and Survival in Mechanically Ventilated Patients With Coronavirus Disease 2019-Related Respiratory Failure. Crit Care Med. 2021 Jul 1;49(7):1026-1037. doi: 10.1097/CCM.0000000000004938. PMID 33595960
- [Background] Mojoli F, Bouhemad B, Mongodi S, Lichtenstein D. Lung Ultrasound for Critically Ill Patients. Am J Respir Crit Care Med. 2019 Mar 15;199(6):701-714. doi: 10.1164/rccm.201802-0236CI. PMID 30372119
- [Background] Jimenez JV, Weirauch AJ, Culter CA, Choi PJ, Hyzy RC. Electrical Impedance Tomography in Acute Respiratory Distress Syndrome Management. Crit Care Med. 2022 Aug 1;50(8):1210-1223. doi: 10.1097/CCM.0000000000005582. Epub 2022 May 23. PMID 35607967
- [Background] He HW, Long Y, Chi Y, Yuan SY, Zhou X, Su LX, Cheng W, Fu F, Zhao ZQ. [Technology specification of bedside hypertonic saline-contrast electrical impedance tomography of lung perfusion and clinical application]. Zhonghua Yi Xue Za Zhi. 2021 Apr 20;101(15):1097-1101. doi: 10.3760/cma.j.cn112137-20200926-02723. Chinese. PMID 33878839
- [Background] He H, Chi Y, Long Y, Yuan S, Zhang R, Frerichs I, Moller K, Fu F, Zhao Z. Bedside Evaluation of Pulmonary Embolism by Saline Contrast Electrical Impedance Tomography Method: A Prospective Observational Study. Am J Respir Crit Care Med. 2020 Nov 15;202(10):1464-1468. doi: 10.1164/rccm.202005-1780LE. No abstract available. PMID 32585116
- [Background] He H, Chi Y, Long Y, Yuan S, Frerichs I, Moller K, Fu F, Zhao Z. Influence of overdistension/recruitment induced by high positive end-expiratory pressure on ventilation-perfusion matching assessed by electrical impedance tomography with saline bolus. Crit Care. 2020 Sep 29;24(1):586. doi: 10.1186/s13054-020-03301-x. PMID 32993811
- [Background] Spinelli E, Kircher M, Stender B, Ottaviani I, Basile MC, Marongiu I, Colussi G, Grasselli G, Pesenti A, Mauri T. Unmatched ventilation and perfusion measured by electrical impedance tomography predicts the outcome of ARDS. Crit Care. 2021 Jun 3;25(1):192. doi: 10.1186/s13054-021-03615-4. PMID 34082795
- [Background] Zarantonello F, Andreatta G, Sella N, Navalesi P. Prone Position and Lung Ventilation and Perfusion Matching in Acute Respiratory Failure due to COVID-19. Am J Respir Crit Care Med. 2020 Jul 15;202(2):278-279. doi: 10.1164/rccm.202003-0775IM. No abstract available. PMID 32437251
- [Derived] Wang R, Wang W, Tang X, Qi Z, Li T, Liu Y, Li H, Yan J, Yang H, Lyu W, Li Z, Sun B, Gan G. Association between ventilation-perfusion matching improvement during initial prone positioning and ICU mortality in patients with moderate to severe ARDS: a prospective two-center study. Ann Intensive Care. 2025 May 21;15(1):69. doi: 10.1186/s13613-025-01489-1. PMID 40394400